CLINICAL TRIAL: NCT04647292
Title: European Blood Pressure Intensive Control After Stroke - Pilot Trial
Brief Title: European Blood Pressure Intensive Control After Stroke
Acronym: EPICS-Pilot
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: St Vincent's University Hospital, Ireland (Other); Cork University Hospital (Other); Tallaght University Hospital (Other); HRB Stroke Trials Network Ireland (Unknown); National University of Ireland, Galway, Ireland (Other); Mater Misericordiae University Hospital (Other); St. James's Hospital, Ireland (Other); Connolly Hospital Blanchardstown (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7580
Record Dates: First submitted 2020-11-20; First posted 2020-11-30 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: ischemic stroke; transient ischemic attack; blood pressure; hypertension; recurrence; prognosis; prevention; randomized control trial; myocardial infarction; vascular events
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Hypertension; Recurrence; Myocardial Infarction | interventions — Antihypertensive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Blood Pressure Measurement, Telemonitoring and Medication titration (Experimental): Medication titration to guideline SBP <130mmHg
  Interventions: Other: anti-hypertensive, home blood pressure measurement, telemonitoring and medication titration
- Control Group: Standard of Care Blood Pressure Management (Active Comparator): Standard of Care Management by GP/physician to SBP <130mmHg by current European Stroke Organisation, American Stroke Association and UK NICE guidelines
  Interventions: Other: Standard of Care Blood Pressure Management with Antihypertensives

INTERVENTIONS:
Other: anti-hypertensive, home blood pressure measurement, telemonitoring and medication titration — A medication algorithm based on the SPRINT trial protocol will be provided for patients in the home blood pressure measurement arm. The final choice and dose of antihypertensive treatment(s) will be at the discretion of the treating clinicians. If no contra-indications, indapamide or other thiazide diuretic and/or angiotensin-converting enzyme (ACE) inhibitor (perindopril or other) will be encouraged as initial therapy, with long-acting calcium-channel antagonists (eg.amlodipine) encouraged as third-line therapy.
  Patients will have their home blood pressure monitoring diary reviewed by the study team. If SBP is out of the allocated target range, a prescription to titrate antihypertensive medication will be sent to the patient at least monthly.
  Arms: Home Blood Pressure Measurement, Telemonitoring and Medication titration
Other: Standard of Care Blood Pressure Management with Antihypertensives — Participants in the standard of care arm will receive antihypertensive therapy at the physician's discretion to the same treatment target of SBP <130mmHg.
  Arms: Control Group: Standard of Care Blood Pressure Management

SUMMARY:
Stroke is the third most common cause of death worldwide and the leading cause of disability. High blood pressure is an important risk factor for stroke. Lowering a person's blood pressure reduces the risk of future stroke or heart attack, and current guidelines recommend treatment to a target of <130mmHg for secondary prevention.

Home blood pressure measurement and telemonitoring are acceptable to patients, but there is uncertainty over the use of out of office blood pressure measurements in stroke patients in guidelines.

This is a study designed to establish the feasibility of a larger clinical trial, comparing home blood pressure monitoring, telemonitoring and medication titration with standard care. The study hypothesis is that home BP measurement and telemonitoring with medication titration may lead to improved BP control compared to standard of care clinical practice.

DETAILED DESCRIPTION:
Background:

Stroke is the third leading cause of global death, the leading cause of acquired disability and contributes substantially to dementia, cognitive decline, and healthcare costs. Global epidemiological studies such as INTERSTROKE and the Global Burden of Disease study estimated that hypertension is the leading modifiable risk factor for stroke, with a population attributable risk of approximately 50%. Recurrent vascular events (stroke, coronary events, vascular death) cause significant morbidity in ischaemic stroke survivors, affecting approximately 30% at 5 years.

High rates of failure to achieve guideline BP targets (<130mmHg) are reported in clinical practice for patients following ischaemic stroke or TIA. Home blood pressure measurement and telemonitoring is recognised as acceptable to patients from previous studies, and some trials have noted a significant reduction in BP at 12 months. The latest ESO guidelines note continued uncertainty over the use of out-of-office blood pressure measurements for adult patients with ischaemic stroke or TIA due to insufficient data.

This trial will recruit patients with recent stroke/TIA events with systolic BP ≥140 mmHg and randomise them to standard of care or home BP monitoring with telemonitoring and medication titration. The study hypothesis is that home BP measurement and telemonitoring with medication titration may lead to improved BP control compared to standard of care clinical practice.

Aim:

The aim is to conduct an initial pilot randomised trial in Ireland and European centres involved in the European Stroke Organisation Trials Alliance. This feasibility study will assess key design aspects and establish trial governance, data management, and procedures in preparation for a larger definitive trial.

Methods:

Design: Prospective, open-label, blinded endpoint assessed (PROBE) randomised, parallel group pilot/feasibility clinical trial, comparing BP patient self-measurement and telemonitoring with office-based monitoring (standard of care) for improved BP control after ischaemic stroke/TIA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40
2. Ischaemic stroke1, high-risk TIA, proven by imaging (brain CT/MRI)
3. Living at home and independent (walking without the aid of another person, but may have some help for daily activities)
4. SBP≥140mmHg at entry (average of 2 measures, seated, in the same arm, after resting alone in office for 10 minutes)
5. Qualifying event between 30 days and 1 year of randomisation
6. Glomerular filtration rate (eGFR) greater than or equal to 50ml/min/m2 (within 3 months of randomisation)
7. Medically-stable and capable of participating in a randomised trial, including home BP measures, in the opinion of the study physician
8. Willing to provide informed consent (no surrogate consent will apply)

Exclusion Criteria:

1. SBP <110mmHg after 3 minutes of standing or other contra-indication to intensive SBP lowering in opinion of treating clinician (eg. Orthostatic symptoms, syncope or pre syncope, recurrent falls)
2. Qualifying stroke due to intracerebral haemorrhage (ICH), cardio-embolism or other defined causes (eg. dissection, endocarditis, other specified)
3. Severe stenosis or occlusion of large cranio-cervical artery (>70% stenosis/occlusion of cervical carotid, vertebral, or Circle of Willis artery)
4. Unlikely to comply with study procedures due to severe or fatal comorbid illness (eg. dementia, active malignancy, severe frailty) or other factor (eg. inability to travel)
5. Pregnancy or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Difference in mean SBP | 12 months (or last trial visit)
  The difference in mean SBP between both groups, at 12 months (or last trial visit)

SECONDARY OUTCOMES:
Proportions of patients assigned to each arm successfully reaching guideline-based target (SBP<130mmHg) at end of trial visit | 12 months (or last trial visit)
Time in guideline-based target range | 12 months (or last trial visit)
  Proportion of SBP measures <130 during trial participation
Time taken to reach target | 12 months (or last trial visit)
  Time taken to reach target SBP<130mmHg
Difference in mean diastolic blood pressure (DBP) between groups | 12 months (or last trial visit)
Change in SBP/DBP from baseline to end-of-trial | 12 months (or last trial visit)
Time to first composite major adverse cardiovascular event (MACE), and to each component of the composite, stratified as fatal, non-fatal and total | 12 months (or last trial visit)
  MACE defined as all recurrent stroke, myocardial infarction, cardiac arrest
All-cause fatality | 12 months (or last trial visit)
Comparison of disability in each intervention arm assessed by modified Rankin score | 12 months (or last trial visit)
  Shift analysis and proportion with no, mild, or moderate disability, Rankin score 0-3
Number of dose-titrations required | 12 months (or last trial visit)
Time required per follow up visit | 12 months (or last trial visit)
Number of patients lost to follow-up | 12 months (or end of trial visit)
Number of serious adverse events | 12 months (or last trial visit)
  Difference in proportion of patients with serious adverse events
Number of pre-specified adverse events | 12 months (or last trial visit)
Change in health related quality of life | 12 months (or last trial visit)
  Change in EQ5D-5L score (5 domains assessed with scores of 1-5 ranking the severity of impairment, with higher scores indicating poorer quality of life) at last follow-up compared with baseline
Change in cognition | 12 months (or last trial visit)
  Change in Montreal cognitive assessment score (range 0-30) at last follow-up compared with baseline score. A lower score indicates greater cognitive impairment.
Qualitative patient feedback obtained via workshops and questionnaires | 12 months (or last trial visit)

OTHER OUTCOMES:
Number of patients who do not complete the study due to tolerability or other issues | 12 months (or end of trial visit)
  Patients who are not retained in the study will give an insight into anticipated retention in the Phase 3 trial and sample size considerations.
Ability of sites to rapidly identify eligible patients from clinics and stroke units | 12 months (or end of trial visit)
  The inclusion of prevalent cases already attending stroke clinics or discharged from stroke units within the last year is an important design feature, aimed to rapidly accrue patients into the trial and thus to maximise the duration of follow-up within the terms allowed by funders. This outcome will be judged on the basis of qualitative feedback from participating sites.
Feasibility of home blood pressure (BP) measures and telemonitoring | 12 months (or end of trial visit)
  This outcome will be judged on the basis of qualitative feedback from participants and the the proportions of participants adhering to the use of home blood pressure diaries.
Compliance with telemonitoring and feasibility of remote (phone) visits | 12 months (or end of trial visit)
  The feasibility of remote (phone) visits will be assessed by the proportion of patients adhering to participation in remote visit consultations
Feasibility of remote BP titration | 12 months (or end of trial visit)
  The feasibility of titration of BP based on prescriptions to pharmacies in response to BP telemonitoring
Barriers to participation of women | 12 months (or end of trial visit)
  Qualitative review to improve the design of a future Phase 3 trial with the aim of reducing barriers to women

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are open to considering requests for collaborative projects.

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903